CLINICAL TRIAL: NCT07047534
Title: Real-time EEG-Triggered Transcranial Magnetic Stimulation Combined With Group Therapy for Adolescents With Depression and Self-Harm Behavior: A Randomized Controlled Trial
Brief Title: EEG-Triggered rTMS and Group Therapy for Adolescents With Depression and Self-Harm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, Yanju Liu, Principal Investigator, The First Hospital of Hebei Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20221425
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2024-06

CONDITIONS: Depression
Keywords: Major Depressive Disorder; Self-Harm Behavior; Adolescent Depression; Transcranial Magnetic Stimulation; Group Therapy
MeSH Terms: conditions — Depression; Depressive Disorder, Major | interventions — Psychotherapy, Group

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real-time EEG-triggered rTMS Alone (Active Comparator): Participants received 20 sessions of real-time EEG-triggered rTMS over 4 weeks (5 sessions/week).
  Interventions: Device: Real-time EEG-triggered Repetitive Transcranial Magnetic Stimulation (rTMS)
- Real-time EEG-triggered rTMS + Group Therapy (Experimental): Participants received identical rTMS (as the control group) plus semi-closed group therapy sessions.
  Interventions: Device: Real-time EEG-triggered Repetitive Transcranial Magnetic Stimulation (rTMS); Behavioral: Group Therapy

INTERVENTIONS:
Device: Real-time EEG-triggered Repetitive Transcranial Magnetic Stimulation (rTMS) — Stimulation target: left dorsolateral prefrontal cortex (DLPFC; F3 electrode position, 10-20 EEG system); Frequency: 10 Hz; Intensity: 110% of resting motor threshold (RMT); Pulse number: 2000 pulses/session (20 trains of 100 pulses, 30-second inter-train interval); EEG triggering: Stimulation pulses synchronized to the peak of the participant's ongoing θ-wave (4-7 Hz) activity. Duration: 20 sessions over 4 weeks.
Behavioral: Group Therapy — Semi-closed group therapy; 10 participants/group, 2 sessions/week, 90 minutes/session for 4 weeks (total 8 sessions). Content included: Sessions 1-2: Emotional recognition and expression training; Sessions 3-4: Cognitive restructuring; Sessions 5-6: Impulse control training; Sessions 7-8: Self-esteem building and future planning.
  Arms: Real-time EEG-triggered rTMS + Group Therapy

SUMMARY:
This randomized controlled trial aims to evaluate the efficacy of real-time EEG-triggered repetitive transcranial magnetic stimulation (rTMS) combined with group therapy versus rTMS alone in adolescents (aged 12-18 years) diagnosed with depression and exhibiting recent self-harm behavior. The primary outcome is the change in depression severity at 4 weeks.

DETAILED DESCRIPTION:
Adolescent depression is a prevalent and severe mood disorder, often comorbid with self-harm behavior, significantly impairing functioning. Repetitive transcranial magnetic stimulation (rTMS) is a non-invasive neuromodulation technique showing promise in depression treatment. Real-time EEG-triggered rTMS (rEEG-TMS) further refines this by synchronizing stimulation with individual neural rhythms, potentially enhancing precision and efficacy. Psychosocial interventions, such as group therapy, are crucial for adolescent mood disorders, offering peer support, emotional regulation skills, and cognitive restructuring. This study investigates whether combining rEEG-TMS with group therapy offers synergistic benefits over rEEG-TMS alone in adolescents with depression and self-harm.

This was a parallel-group randomized controlled trial. A total of 160 inpatients aged 12-18 years with a diagnosis of major depressive disorder (ICD-10 F32) and documented self-harm behavior within 2 weeks prior to enrollment were recruited. Participants were randomized 1:1 to either receive real-time EEG-triggered rTMS alone (control group, n=80) or real-time EEG-triggered rTMS plus group therapy (observation group, n=80). The rTMS intervention consisted of 20 sessions over 4 weeks (5 sessions/week), targeting the left dorsolateral prefrontal cortex (DLPFC) at 10 Hz, 110% of resting motor threshold, with 2000 pulses per session, triggered by the peak of the participant's ongoing θ-wave activity. The group therapy intervention, for the observation group, consisted of 8 semi-closed sessions (2 sessions/week for 4 weeks, 90 minutes/session) covering emotional recognition, cognitive restructuring, impulse control, and self-esteem building. Assessments were conducted at baseline and at 4 weeks post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 12-18 years;
* Diagnosis of major depressive disorder (MDD) according to the International Classification of Diseases, 10th Revision (ICD-10 F32);
* Documented self-harm behavior within 2 weeks prior to enrollment (defined as deliberate self-injury without suicidal intent, e.g., cutting, burning);
* Hamilton Depression Rating Scale (HAMD-24) score ≥17 at baseline;
* Ability to complete self-report measures and participate in group therapy.

Exclusion Criteria:

* Comorbid psychotic disorders (e.g., schizophrenia), bipolar disorder, or autism spectrum disorder;
* History of neurological conditions (e.g., epilepsy, traumatic brain injury);
* Current use of electroconvulsive therapy;
* Refusal to provide informed consent.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 160 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Hamilton Depression Rating Scale (HAMD-24) scores | Baseline and Week 4 (post-intervention)
  The HAMD-24 is a clinician-rated scale to assess the severity of depressive symptoms. Higher scores indicate greater severity of depression. Change is calculated as score at week 4 minus score at baseline.

SECONDARY OUTCOMES:
Change in Hamilton Anxiety Rating Scale (HAMA-14) scores | Baseline and Week 4
  The HAMA-14 is a clinician-rated scale to assess the severity of anxiety symptoms. Higher scores indicate greater severity. Change is calculated as score at week 4 minus score at baseline.
Change in Suicide Probability Scale (SPS) scores | Baseline and Week 4
  The SPS is a self-report measure assessing suicide risk. Scores range from 0-100, with higher scores indicating greater risk. Change is calculated as score at week 4 minus score at baseline.
Change in Modified Self-Harm Inventory (MSHI) scores | Baseline and Week 4
  The MSHI assesses the frequency (0-4) and severity (0-4) of self-harm acts, with a total score ranging from 0-8. Higher scores indicate more severe self-harm behavior. Change is calculated as score at week 4 minus score at baseline.
Change in Event-Related Potential (ERP) P300 Latency | Baseline and Week 4
  P300 latency (measured in milliseconds, ms) recorded during a visual Oddball paradigm at the Cz electrode. Shorter latency generally indicates faster cognitive processing speed. Change is calculated as value at week 4 minus value at baseline.
Change in Event-Related Potential (ERP) P300 Amplitude | Baseline and Week 4
  P300 amplitude (measured in microvolts, μV) recorded during a visual Oddball paradigm at the Cz electrode. Larger amplitude generally indicates greater allocation of neural resources. Change is calculated as value at week 4 minus value at baseline.
Change in Resting-State EEG α (alpha) Power | Baseline and Week 4
  Alpha power (8-12 Hz, measured in μV²) calculated over 3 minutes of eyes-closed resting state EEG. Change is calculated as value at week 4 minus value at baseline.
Change in Resting-State EEG θ (theta) Power | Baseline and Week 4
  Theta power (4-7 Hz, measured in μV²) calculated over 3 minutes of eyes-closed resting state EEG. Change is calculated as value at week 4 minus value at baseline.
Change in Resting-State EEG θ/β (theta/beta) Ratio | Baseline and Week 4
  Theta/beta ratio (beta=13-30 Hz) calculated over 3 minutes of eyes-closed resting state EEG. Change is calculated as value at week 4 minus value at baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Hebei Medical University, Shijiazhuang, Hebei, China

REFERENCES:
- [Derived] Liu H, Liu S, Yu M, Xin B, Liu Y. Real-time EEG-triggered transcranial magnetic stimulation combined with group therapy for adolescents with depression and self-harm behavior: A randomized controlled trial. J Affect Disord. 2026 Jan 1;392:120144. doi: 10.1016/j.jad.2025.120144. Epub 2025 Aug 26. PMID 40876639